CLINICAL TRIAL: NCT00334698
Title: A Randomized, Double Blind, Placebo-controlled, Four Way Cross-over Study to Assess the Effect of a Combination of Cetirizine With Pseudoephedrine Versus Cetirizine Alone on Symptoms Scores and Rhinomanometry in Patients With Allergic Rhinitis Following Pollen Exposure in the Fraunhofer Environmental Challenge Chamber (ECC)
Brief Title: Study to Assess the Effect of a Combination of Cetirizine With Pseudoephedrine Versus Cetirizine Alone on Symptoms in Patients With Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06/02 Nacon ITEM
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2007-05

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Cetirizine; Pseudoephedrine

INTERVENTIONS:
Drug: Cetirizine
Drug: Pseudoephedrine
Drug: Cetirizine with Pseudoephedrine

SUMMARY:
The aim of this study is to assess the efficacy on nasal congestion and other allergic symptoms and the onset of action of an oral combination of cetirizine and pseudoephedrine in comparison to the single substances under controlled pollen exposure in an Environmental Challenge Chamber (ECC).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-55 years.
* Women will be considered for inclusion if they are:

  * Not pregnant, as confirmed by pregnancy test (see flow chart) and not nursing.
  * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
  * Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomized partner, abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication and to continue until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, some IUDs)
* FEV1 > 80% of predicted at screening.
* Absence of any structural nasal abnormalities or nasal polyps on examination, absence of a history of frequent nose bleeding or recent nasal surgery.
* Absence of conditions or factors, which would make the subject unlikely to be able to stay in the Fraunhofer ECC for 6 hours.
* Non smokers or smokers with a history of less than 10 pack years.
* Able and willing to give written informed consent to take part in the study.
* Available to complete all study measurements.
* History of allergic rhinitis to grass pollen and a positive skin prick test for Dactylis glomerata pollen at or within 12 months prior to the screening visit.
* Subject must exhibit a moderate response upon 4000 Dactylis glomerata pollen grains/m3 during 2 hours in the ECC on visit 2.
* Subjects with mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function may be included.

Exclusion Criteria:

* History of a respiratory tract infection and/or exacerbation of asthma within 4 weeks before the screening and during the study.
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures.
* Administration of oral, injectable or dermal corticosteroids within 8 weeks or intranasal and/or inhaled corticosteroids within 4 weeks of the screening visit.
* Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDS), anti-depressant drugs, anti-histamines and anti-asthma, anti-rhinitis or hay fever medication (other than short acting inhaled beta-agonists) for 1 week prior to screening and throughout the course of the study.
* Paracetamol up to 1g per day is permitted for the treatment of minor ailments, e.g. headache.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Known hypersensitivity, allergic reactions or intolerance to cetirizine, pseudoephedrine or any of the other ingredients.
* Subject receiving monoamine oxidase inhibitors or has received these agents in the last two weeks before dosing.
* Subject is undergoing allergen desensitisation therapy.
* There is a risk of non-compliance with study procedures.
* Participation in another clinical trial 30 days prior to enrolment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2006-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change of nasal obstruction symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Norbert Krug, MD, Principal Investigator — Fraunhofer Institute of Toxikology and Experimental Medicine
Locations (1):
- Fraunhofer-Institute of Toxicology and Experimental Medicine, Hanover, Germany